CLINICAL TRIAL: NCT01282307
Title: Meaningful Change With the Method Guided Self-Determination - a Randomised Controlled Study for Patients Diagnosed With Schizophrenia.
Brief Title: Improving Insight in Patients Diagnosed With Schizophrenia
Acronym: GEBRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aalborg Psychiatric Hospital (Other)
Responsible Party: Principal Investigator, Rikke Jørgensen, MSN ResearchNurse, PhD.Student, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20070070
Record Dates: First submitted 2010-11-19; First posted 2011-01-24 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Schizophrenia
Keywords: Guided Self-Determination; Improving insight; Autonomy-supportive problem solving intervention; Evaluate the effects of the method Guided Self-Determination; Improving insight in patients diagnosed with schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Method Guided Self-Determination (Experimental): The Method Guided Self-Determination consists of 21 worksheets designed to guide patient and mental health professionals through autonomy-supportive problem solving. The worksheets are filled in by the patient before and between conversations with their community nurse over 10 sessions, approximately 1 hour a session.
  Interventions: Behavioral: Guided Self-Determination GSD
- Treatment as usual (No Intervention)

INTERVENTIONS:
Behavioral: Guided Self-Determination GSD — The method GSD consists of 21 worksheets designed to guide patient and mental health professionals through autonomy-supportive problem solving. The worksheets are filled in by the patient before and between conversations with their community nurse over 10 sessions, approximately 1 hour a session.
  Arms: Method Guided Self-Determination

SUMMARY:
Background:

Rehospitalisation and discontinued treatment are common among patients with schizophrenia and is often associated with lack of insight into the illness. Improving patients' insight has been attempted through psychoeducation and standard treatment but without any considerable change. A newly developed method, Guided Self-Determination (GSD), originally developed and proved effective in difficult diabetes care has been adjusted to patients with schizophrenia. A qualitative evaluation of GSD has shown a positive influence on patients' insight into the illness.

Aim and hypotheses: The aim of the study is to evaluate the effects of the method GSD in the care of patients with schizophrenia compared to treatment as usual. The following hypotheses will be tested:

The method GSD will improve: Cognitive and clinical insight in patients, various domains of recovery, patients' self-esteem, psychopathology and social functioning.

Material and method:

The study design is a randomised controlled trial. The participants are diagnosed with schizophrenia and schizoaffective disorder, receiving treatment in 3 Assertive Outreach Teams and 3 Psychosis Teams in Region North. Participants complete four self-rating questionnaires, a demographic data sheet, an interview concerning psychopathology and an assessment of social functioning at baseline, and after 3, 6, and 12 month. All assessments will be conducted by the investigator, except for the assessment of social functioning, that will be measures by community nurses. Intervention with the method GSD will also be conducted by the community nurses but under supervision from the investigator. Fifty patients are randomly assigned to immediate receipt of individual training with the method GSD (intervention group) and 50 to a 12-month waiting list for individual training with the method GSD (control group).

Perspectives:

In mental health nursing practice in Denmark there is no tradition for empirical research as the basis of psychiatric nursing - unverified theories or general empirical consensus of good clinical practice are often the foundation of psychiatric nursing. If the method GSD proves effective in the care of patients with schizophrenia, this study contributes to an evidence based nursing intervention, which is ready for further research on implementation in mental health nursing practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient's hospital record meeting the criteria for schizophrenia according to ICD-10 F.20.0-9 or schizoaffective disorder according to ICD-10 F.25.0-9
* Age 18 - 70 years at the time of inclusion
* Ability to understand, speak and write Danish - assessed by the community nurse
* Informed written consent
* receiving treatment in an assertive outreach team or psychosis team in region north in Denmark

Exclusion Criteria:

* Previous participation with the method GSD
* Patients who are mentally handicapped or diagnosed with any kind of dementia or an organic brain disease according to their hospital record
* In need of an interpreter to understand, speak and write Danish
* Withdrawal of informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
changes in cognitive insight over time | baseline, 3,6 and 12 month
  Cognitive insight is measured by the selvrating questionnaire Beck Cognitive Insight Scale (BCIS).

SECONDARY OUTCOMES:
Changes in Clinical insight over time | baseline, 3,6,12 month
  Clinical insight is measured by the self-rating questionnaire "Birchwood Insight Scale"
changes in various domains of recovery over time | baseline, 3,6,12 month
  recovery is measured by the self-rating questionnaire "Recovery Assessment Scale"
changes in self-esteem over time | baseline, 3,6,12 month
  self-esteem is measured by the self-rating questionnaire "Rosenberg self-esteem scale"
changes in psychopathology over time | baseline, 3,6,12 month
  Psychopathology is measured by the PANSS - "Positive and Negative Symptom Scale"
changes of social function over time | baseline, 3,6,12 month
  Social function is measured by GAF - "Global Assessment Scale"
Therapeutic relationship | 12 month
  Therapeutic relationship is measured by STAR - "Scale to assess Therapeutic Relationship in Community Mental Health Care" patient version
Therapeutic relationship | 12 month
  Therapeutic relationship is measured by HAS - "Helping Alliance Scale"

CONTACTS AND LOCATIONS:
Overall Officials: Rikke Jørgensen, MSN, Principal Investigator — Unit for Psychiatric Research, Aalborg Psychiatric Hospital
Locations (1):
- Psychiatry in Region North Jutland, Aalborg, North Jutland, Denmark

REFERENCES:
- [Derived] Jorgensen R, Licht RW, Lysaker PH, Munk-Jorgensen P, Buck KD, Jensen SO, Hansson L, Zoffmann V. Effects on cognitive and clinical insight with the use of Guided Self-Determination in outpatients with schizophrenia: A randomized open trial. Eur Psychiatry. 2015 Jul;30(5):655-63. doi: 10.1016/j.eurpsy.2014.12.007. Epub 2015 Jan 16. PMID 25601635